CLINICAL TRIAL: NCT03354637
Title: A Randomized, Double-Blind, Vehicle-Controlled Multicenter Study to Evaluate the Safety, Tolerability and Efficacy of ATI-50002 Topical Solution Administered Twice-Daily for 6 Months in Adolescents and Adult Subjects With Stable Patchy Alopecia Areata With Optional Long-Term Open-Label Extension
Brief Title: A Study of ATI-50002 Topical Solution for the Treatment of Alopecia Areata
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The double-blind primary endpoint was not met. Open Label Extension period halted as a result.
Sponsor: Aclaris Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ATI-50002-AA-201
Record Dates: First submitted 2017-11-16; First posted 2017-11-28 (Actual); Results first posted 2020-06-05 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-05

CONDITIONS: Alopecia Areata
MeSH Terms: conditions — Alopecia Areata

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ATI-50002 high dose Topical Solution (Active Comparator): High dose active
  Interventions: Drug: ATI-50002 high dose
- ATI-50002 low dose Topical Solution (Active Comparator): low dose active
  Interventions: Drug: ATI-50002 low dose
- Vehicle Topical Solution (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ATI-50002 high dose — Topical solution
  Arms: ATI-50002 high dose Topical Solution
Drug: ATI-50002 low dose — Topical solution
  Arms: ATI-50002 low dose Topical Solution
Drug: Placebo — Topical solution
  Arms: Vehicle Topical Solution

SUMMARY:
Primary:

• To assess safety, tolerability and efficacy of 2 dose strengths of ATI-50002 Topical Solution, compared to vehicle in subjects with alopecia areata (AA)

Secondary:

• To evaluate key clinical outcome assessments

DETAILED DESCRIPTION:
Primary:

• To assess safety, tolerability and efficacy of 2 dose strengths of ATI-50002 Topical Solution, compared to vehicle in subjects with alopecia areata (AA)

Secondary:

• To evaluate key clinical outcome assessments

ELIGIBILITY:
Inclusion Criteria:

1. Have a clinical diagnosis of stable patchy alopecia areata (AA) defined as no current areas of spontaneous regrowth.
2. Have a Severity of Alopecia Tool (SALT) score of at least 15% up to 95% total scalp hair loss determined by the study investigator at baseline.
3. Have a duration of the current episode of scalp hair loss of a minimum of 6 months and a maximum of 12 years.
4. If a woman of childbearing potential (WOCBP), must have a negative serum pregnancy test at Screening (Visit 1) and a negative urine pregnancy test at Baseline (Visit 2) and agree to: use a highly effective method of birth control for the duration of the study; not be planning a pregnancy during the study duration and use contraception for 30 days after last application of study medication.

Exclusion Criteria:

1. Females who are nursing, pregnant, or planning to become pregnant for the duration of the study and up to 30 days after the last application of study medication.
2. Diffuse alopecia areata.
3. Concomitant hair loss disorder (by history or physical exam) such as androgenetic alopecia or scarring alopecia (e.g., cicatricial alopecia, frontal fibrosing alopecia, etc.).
4. Active skin disease on the scalp (such as psoriasis or seborrheic dermatitis) or a history of skin disease on the scalp that in the opinion of the investigator would interfere with the study assessments of efficacy or safety.
5. Active scalp trauma or other condition affecting the scalp that, in the investigator's opinion, may affect the course of AA or interfere with the study conduct or evaluations.
6. The presence of a permanent or difficult to remove hairpiece or wig that will, in the opinion of the investigator, interfere with study assessments if not removed at each visit.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2017-11-29 (Actual); Primary Completion 2019-04-18 (Actual); Study Completion 2019-09-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (21):
- United States (21):
  - Aclaris Investigator Site, Encinitas, California
  - Aclaris Investigator Site, Laguna Hills, California
  - Aclaris Investigator Site, Redwood City, California
  - Aclaris Investigator Site, Washington D.C., District of Columbia
  - Aclaris Investigator Site, Boynton Beach, Florida
  - Aclaris Investigator Site, Miami, Florida
  - Aclaris Investigator Site, Boston, Massachusetts
  - Aclaris Investigator Site, Clinton Township, Michigan
  - Aclaris Investigator Site, Warren, Michigan
  - Aclaris Investigator Site, Fridley, Minnesota
  - Aclaris Investigator Site, Minneapolis, Minnesota
  - Aclaris Investigator Site, Omaha, Nebraska
  - Aclaris Investigator Site, New York, New York
  - Aclaris Investigator Site, Durham, North Carolina
  - Aclaris Investigator Site, Winston-Salem, North Carolina
  - Aclaris Investigator Site, Portland, Oregon
  - Aclaris Investigator Site, Fort Washington, Pennsylvania
  - Aclaris Investigator Site, Knoxville, Tennessee
  - Aclaris Investigator Site, Nashville, Tennessee
  - Aclaris Investigator Site, Austin, Texas
  - Aclaris Investigator Site, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Vehicle Topical Solution: Vehicle Topical Solution applied twice daily.
- ATI-50002 0.12% Topical Solution: ATI-50002 0.12% Topical Solution applied twice daily.
- ATI-50002 0.46% Topical Solution: ATI-50002 0.46% Topical Solution applied twice daily.
Period: Double-blind Period
Arm/Group | Vehicle Topical Solution | ATI-50002 0.12% Topical Solution | ATI-50002 0.46% Topical Solution
Started | 43 | 44 | 42
Completed | 26 | 31 | 35
Not Completed | 17 | 13 | 7
Not completed — Protocol Violation | 2 | 0 | 0
Not completed — Adverse Event | 1 | 2 | 0
Not completed — Lost to Follow-up | 3 | 4 | 3
Not completed — Withdrawal by Subject | 10 | 6 | 4
Not completed — Incomplete Efficacy Data Collection | 1 | 1 | 0
Period: Open Label Extension
Arm/Group | Vehicle Topical Solution | ATI-50002 0.12% Topical Solution | ATI-50002 0.46% Topical Solution
Started (Subjects entering the Open Label Extension period all received ATI-50002 0.46% Topical Solution.) | 0 | 0 | 61
Completed | 0 | 0 | 33
Not Completed | 0 | 0 | 28
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 5
Not completed — Study Terminated by Sponsor | 0 | 0 | 17
Not completed — Subject Noncompliance | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vehicle Topical Solution | ATI-50002 0.12% Topical Solution | ATI-50002 0.46% Topical Solution | Total
Number analyzed (Participants) | 43 | 44 | 42 | 129
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 0 | 2 | 5
  Between 18 and 65 years | 36 | 40 | 37 | 113
  >=65 years | 4 | 4 | 3 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.0 (16.58) | 42.1 (13.92) | 40.5 (14.99) | 41.5 (15.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 13 | 18 | 46
  Male | 28 | 31 | 24 | 83
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 4 | 7 | 19
  Not Hispanic or Latino | 23 | 26 | 23 | 72
  Unknown or Not Reported | 12 | 14 | 12 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 11 | 10 | 7 | 28
  White | 32 | 29 | 31 | 92
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 43 | 43 | 43 | 129
Fitzpatrick Skin Type [Count of Participants; unit: Participants]
  I - Always Burns | 2 | 3 | 2 | 7
  II - Burns Easily | 12 | 16 | 14 | 42
  III - Burns Moderately | 13 | 9 | 9 | 31
  IV - Burns Minimally | 6 | 6 | 8 | 20
  V - Rarely Burns | 6 | 7 | 6 | 19
  VI - Never Burns | 4 | 3 | 3 | 10
Duration of Current Episode of Alopecia Areata [Mean (Standard Deviation); unit: weeks] | 127.8 (104.13) | 160.7 (140.67) | 156.3 (140.95) | 148.3 (129.55)
Duration of Alopecia Areata [Mean (Standard Deviation); unit: years] | 6.9 (7.92) | 12.9 (12.25) | 9.9 (10.43) | 9.9 (10.59)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in the Severity of Alopecia Tool Score at Week 24
Description: The Severity of Alopecia Tool (SALT) score is a physician administered scale measuring the amount of scalp without any terminal hair assessed by the investigator at Baseline, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 24. Possible scores range from 0 (no scalp hair loss) to 100 (complete scalp hair loss). A negative change in the SALT score over time represents hair regrowth. The primary efficacy variable was the percent change from baseline in SALT score at Week 24. This was calculated as the mean of the changes from Baseline (Visit 2) SALT score to Week 24 (Visit 10) SALT score, divided by Baseline SALT score and expressed as a percentage.
Time Frame: Baseline - Week 24
Population: This primary analysis utilized the SALT score with imputation for last observation carried forward (LOCF) and was based on the intent-to-treat population.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Vehicle Topical Solution | ATI-50002 0.12% Topical Solution | ATI-50002 0.46% Topical Solution
Number analyzed (Participants) | 43 | 44 | 42
score on a scale | -18.54 (4.705) | -4.66 (4.707) | -9.22 (4.784)
Statistical Analysis 1: Comparison: Vehicle Topical Solution vs ATI-50002 0.12% Topical Solution; Since this was the first multicenter study evaluating the effect of ATI-50002 Topical Solution in subjects with stable patchy alopecia areata, the sample size was based upon feasibility issues rather than a formal power calculation. Planned data from 120 subjects, utilizing LOCF for missing data, provides 80% power to detect a 24-point difference in percent change from baseline in SALT score between any two treatment groups. This power computation is based upon assumed standard deviation of 38%; Test type: Superiority; p = 0.038, Mixed Models Analysis — All statistical testing was two-sided and performed using a significance (alpha) level of 0.05; Mean Difference (Final Values) = 13.88, 95% CI 2-sided [0.77 to 27.00], Standard Error of Mean 4.707
Statistical Analysis 2: Comparison: Vehicle Topical Solution vs ATI-50002 0.46% Topical Solution; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.166, Mixed Models Analysis — All statistical testing was two-sided and performed using a significance (alpha) level of 0.05; Mean Difference (Final Values) = 9.32, 95% CI 2-sided [-3.90 to 22.55], Standard Error of Mean 4.784

2. Secondary Outcome: Percent Change From Baseline in the Alopecia Density and Extent Score at Week 24
Description: The Alopecia Density and Extent (ALODEX) score is a measurement of the amount of scalp with terminal hair loss assessed by the investigator at Baseline, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 24. ALODEX breaks the scalp up into a grid of 1% scalp surface areas and assigns density rating in each area on a 10 point scale of hair loss (0= no hair loss to 10 = complete baldness). Summation of scores from each 1% scalp surface area provides an overall score which may range from 0 (no scalp hair loss) to 100 (complete baldness). A negative change in the ALODEX score over time represents hair regrowth.
Time Frame: Baseline - Week 24
Population: Intent-to-treat population using LOCF to address missing data.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Vehicle Topical Solution | ATI-50002 0.12% Topical Solution | ATI-50002 0.46% Topical Solution
Number analyzed (Participants) | 43 | 44 | 42
score on a scale | -14.75 (4.508) | -8.15 (4.511) | -11.52 (4.584)
Statistical Analysis 1: Comparison: Vehicle Topical Solution vs ATI-50002 0.12% Topical Solution; Test type: Superiority; p = 0.302, Mixed Models Analysis; Mean Difference (Final Values) = 6.60, 95% CI 2-sided [-5.97 to 19.17], Standard Error of Mean 4.511
Statistical Analysis 2: Comparison: Vehicle Topical Solution vs ATI-50002 0.46% Topical Solution; Test type: Superiority; p = 0.616, Mixed Models Analysis; Mean Difference (Final Values) = 3.23, 95% CI 2-sided [-9.44 to 15.90], Standard Error of Mean 4.584

3. Secondary Outcome: Mean Change From Baseline in Severity of Alopecia Tool Score at Week 24
Description: The Severity of Alopecia Tool (SALT) score is a physician administered scale measuring the amount of scalp without any terminal hair. Possible scores range from 0 (no scalp hair loss) to 100 (complete scalp hair loss). A negative change in the SALT score over time represents hair regrowth.
Time Frame: Baseline - Week 24
Population: Intent-to-treat population using LOCF to address missing data.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Vehicle Topical Solution | ATI-50002 0.12% Topical Solution | ATI-50002 0.46% Topical Solution
Number analyzed (Participants) | 43 | 44 | 42
score on a scale | -6.47 (2.071) | -1.95 (2.074) | -2.94 (2.107)
Statistical Analysis 1: Comparison: Vehicle Topical Solution vs ATI-50002 0.12% Topical Solution; Test type: Superiority; p = 0.125, Mixed Models Analysis; Mean Difference (Final Values) = 4.52, 95% CI 2-sided [-1.26 to 10.30], Standard Error of Mean 2.074
Statistical Analysis 2: Comparison: Vehicle Topical Solution vs ATI-50002 0.46% Topical Solution; Test type: Superiority; p = 0.234, Mixed Models Analysis; Mean Difference (Final Values) = 3.53, 95% CI 2-sided [-2.30 to 9.36], Standard Error of Mean 2.107

4. Secondary Outcome: Mean Change From Baseline in Alopecia Density and Extent Score at Week 24
Description: as for outcome 2
Time Frame: Baseline - Week 24
Population: Intent-to-treat population using LOCF to address missing data.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Vehicle Topical Solution | ATI-50002 0.12% Topical Solution | ATI-50002 0.46% Topical Solution
Number analyzed (Participants) | 43 | 44 | 42
score on a scale | -4.91 (2.129) | -3.36 (2.131) | -4.98 (2.165)
Statistical Analysis 1: Comparison: Vehicle Topical Solution vs ATI-50002 0.12% Topical Solution; Test type: Superiority; p = 0.607, Mixed Models Analysis; Mean Difference (Final Values) = 1.55, 95% CI 2-sided [-4.39 to 7.49], Standard Error of Mean 2.131
Statistical Analysis 2: Comparison: Vehicle Topical Solution vs ATI-50002 0.46% Topical Solution; Test type: Superiority; p = 0.981, Mixed Models Analysis; Mean Difference (Final Values) = -0.07, 95% CI 2-sided [-6.06 to 5.92], Standard Error of Mean 2.165

5. Secondary Outcome: Proportion of Subjects Achieving ≥50% Hair Regrowth Based on Severity of Alopecia Tool Scores at Week 24
Description: A summary of the proportion of subjects in each treatment arm achieving ≥50% hair regrowth compared with baseline using Severity of Alopecia Tool scores at Week 24 is presented.
Time Frame: Baseline - Week 24
Population: Intent-to-treat population using LOCF to address missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle Topical Solution | ATI-50002 0.12% Topical Solution | ATI-50002 0.46% Topical Solution
Number analyzed (Participants) | 43 | 44 | 42
Participants | 5 | 7 | 8
Statistical Analysis 1: Comparison: Vehicle Topical Solution vs ATI-50002 0.12% Topical Solution; Test type: Superiority; p = 0.620, Mixed Models Analysis; Odds Ratio (OR) = 1.4, 95% CI 2-sided [0.4 to 4.6]
Statistical Analysis 2: Comparison: Vehicle Topical Solution vs ATI-50002 0.46% Topical Solution; Test type: Superiority; p = 0.366, Mixed Models Analysis; Odds Ratio (OR) = 1.7, 95% CI 2-sided [0.5 to 5.8]

6. Secondary Outcome: Proportion of Subjects Achieving ≥50% Hair Regrowth Based on Alopecia Density and Extent Scores at Week 24
Description: A summary of the proportion of subjects in each treatment arm achieving ≥50% hair regrowth compared with baseline using Alopecia Density and Extent scores at Week 24 is presented.
Time Frame: Baseline - Week 24
Population: Intent-to-treat population using LOCF to address missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle Topical Solution | ATI-50002 0.12% Topical Solution | ATI-50002 0.46% Topical Solution
Number analyzed (Participants) | 43 | 44 | 42
Participants | 6 | 8 | 8
Statistical Analysis 1: Comparison: Vehicle Topical Solution vs ATI-50002 0.12% Topical Solution; Test type: Superiority; p = 0.157, Mixed Models Analysis; Odds Ratio (OR) = 0.1, 95% CI 2-sided [0.0 to 2.3]
Statistical Analysis 2: Comparison: Vehicle Topical Solution vs ATI-50002 0.46% Topical Solution; Test type: Superiority; p = 0.353, Mixed Models Analysis; Odds Ratio (OR) = 0.4, 95% CI 2-sided [0.1 to 2.8]

7. Secondary Outcome: Proportion of Subjects With ≥2 Point Improvement in Scalp Patient Reported Outcome for Target Patch at Week 24
Description: The Scalp Patient Reported Outcome for Target Patch assesses the appearance of the subject's target patch (identified by the subject as his or her most bothersome area of scalp hair loss at Baseline) and was completed by subjects at Baseline, Week 4, Week 12, and Week 24. The assessment has a recall period of "right now" and includes a five-point VRS ranging from "Full hair, scalp of the target patch completely covered with hair" to "no hair, scalp of the target patch completely exposed." The instrument produces a score of 1 to 5, with lower scores indicating more hair covering the subject's target patch. A summary of the proportion of subjects with ≥2 point improvement in Subject Target Patch assessment at Week 24 compared to baseline is presented.
Time Frame: Baseline - Week 24
Population: Intent-to-treat population using LOCF to address missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle Topical Solution | ATI-50002 0.12% Topical Solution | ATI-50002 0.46% Topical Solution
Number analyzed (Participants) | 43 | 44 | 42
Participants | 6 | 8 | 9
Statistical Analysis 1: Comparison: Vehicle Topical Solution vs ATI-50002 0.12% Topical Solution; Test type: Superiority; p = 0.333, Mixed Models Analysis; Odds Ratio (OR) = 1.7, 95% CI 2-sided [0.6 to 5.4]
Statistical Analysis 2: Comparison: Vehicle Topical Solution vs ATI-50002 0.46% Topical Solution; Test type: Superiority; p = 0.388, Mixed Models Analysis; Odds Ratio (OR) = 1.7, 95% CI 2-sided [0.5 to 5.2]

8. Secondary Outcome: Proportion of Subjects With ≥1 Point Improvement in Scalp Patient Reported Outcome for Entire Scalp at Week 24
Description: The Scalp Patient Reported Outcome for Entire Scalp assesses the appearance of the subject's whole scalp and was completed by subjects at Baseline, Week 4, Week 12, and Week 24. The assessment has a recall period of "right now" and includes a five-point VRS ranging from "Full hair, whole scalp completely covered with hair" to "no hair, whole scalp completely exposed." The instrument produces a score of 1 to 5, with lower scores indicating more hair covering the subject's target patch. A summary of the proportion of subjects with ≥1 point improvement in Subject Entire Scalp assessment at Week 24 compared to baseline is presented.
Time Frame: Baseline - Week 24
Population: Intent-to-treat population using LOCF to address missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle Topical Solution | ATI-50002 0.12% Topical Solution | ATI-50002 0.46% Topical Solution
Number analyzed (Participants) | 43 | 44 | 42
Participants | 13 | 10 | 9
Statistical Analysis 1: Comparison: Vehicle Topical Solution vs ATI-50002 0.12% Topical Solution; Test type: Superiority; p = 0.435, Mixed Models Analysis; Odds Ratio (OR) = 0.7, 95% CI 2-sided [0.3 to 1.8]
Statistical Analysis 2: Comparison: Vehicle Topical Solution vs ATI-50002 0.46% Topical Solution; Test type: Superiority; p = 0.370, Mixed Models Analysis; Odds Ratio (OR) = 0.6, 95% CI 2-sided [0.2 to 1.7]

9. Secondary Outcome: Proportion of Subjects With ≥2-Point Improvement in Scalp Clinician Reported Outcome for Target Patch at Week 24
Description: The Scalp Clinician Reported Outcome for Target Patch provides the investigator's assessment of the appearance of the subject's target patch (identified by the subject as his or her most bothersome area of scalp hair loss at Baseline) and was completed by investigators at Baseline, Week 4, Week 12, and Week 24. The assessment has a recall period of "right now" and includes a five-point VRS ranging from "Full hair, scalp of the target patch completely covered with hair" to "no hair, scalp of the target patch completely exposed." The instrument produces a score of 1 to 5, with lower scores indicating more hair covering the subject's target patch. A summary of the proportion of subjects with ≥2 point improvement in Clinician Target Patch assessment at Week 24 compared to baseline is presented.
Time Frame: Baseline - Week 24
Population: Intent-to-treat population using LOCF to address missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle Topical Solution | ATI-50002 0.12% Topical Solution | ATI-50002 0.46% Topical Solution
Number analyzed (Participants) | 43 | 44 | 42
Participants | 6 | 10 | 9
Statistical Analysis 1: Comparison: Vehicle Topical Solution vs ATI-50002 0.12% Topical Solution; Test type: Superiority; p = 0.333, Mixed Models Analysis; Odds Ratio (OR) = 1.7, 95% CI 2-sided [0.6 to 5.4]
Statistical Analysis 2: Comparison: Vehicle Topical Solution vs ATI-50002 0.46% Topical Solution; Test type: Superiority; p = 0.388, Mixed Models Analysis; Odds Ratio (OR) = 1.7, 95% CI 2-sided [0.5 to 5.2]

10. Secondary Outcome: Change From Baseline in Scalp Clinician Reported Outcome for Entire Scalp at Week 24
Description: The Scalp Clinician Reported Outcome for Entire Scalp assesses the appearance of the subject's whole scalp and was completed by investigators at Baseline, Week 4, Week 12, and Week 24. The assessment has a recall period of "right now" and includes a five-point VRS ranging from "Full hair, whole scalp completely covered with hair" to "no hair, whole scalp completely exposed." The instrument produces a score of 1 to 5, with lower scores indicating more hair covering the subject's target patch. Change status is categorized as 'Better by x points' when the score decreases from baseline by x points, and as 'Worse by x points' when the score increases by x points.
Time Frame: Baseline - Week 24
Population: Intent-to-treat population using LOCF to address missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle Topical Solution | ATI-50002 0.12% Topical Solution | ATI-50002 0.46% Topical Solution
Number analyzed (Participants) | 43 | 44 | 42
Participants
  Better by 4 points | 0 | 0 | 0
  Better by 3 points | 0 | 0 | 1
  Better by 2 points | 1 | 2 | 2
  Better by 1 points | 11 | 9 | 8
  No change | 27 | 27 | 23
  Worse by 1 point | 4 | 5 | 7
  Worse by 2 point | 0 | 1 | 1
  Worse by 3 point | 0 | 0 | 0
  Worse by 4 point | 0 | 0 | 0
Statistical Analysis 1: Comparison: Vehicle Topical Solution vs ATI-50002 0.12% Topical Solution; Test type: Superiority; p = 0.505, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Vehicle Topical Solution vs ATI-50002 0.46% Topical Solution; Test type: Superiority; p = 0.359, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Change From Baseline in the Physician Global Impression of Severity (PhGIS) of Patchy Alopecia Areata at Week 24
Description: The Physician Global Impression of Severity (PhGIS) is a 5-point descriptive scale completed by investigators at Baseline, Week 4, Week 12, and Week 24 and is used to capture the investigator's assessment of the subject's disease severity at a particular timepoint. Scores of 1 to 5 are assigned to responses Mild to Extremely Severe, respectively. Change status is categorized as 'Better by x points' when the score decreases from baseline by x points, and as 'Worse by x points' when the score increases by x points.
Time Frame: Baseline - Week 24
Population: Intent-to-treat population using LOCF to address missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle Topical Solution | ATI-50002 0.12% Topical Solution | ATI-50002 0.46% Topical Solution
Number analyzed (Participants) | 43 | 44 | 42
Participants
  Better by 4 points | 0 | 0 | 0
  Better by 3 points | 0 | 0 | 0
  Better by 2 points | 5 | 4 | 4
  Better by 1 point | 9 | 10 | 12
  No change | 27 | 26 | 19
  Worse by 1 point | 1 | 3 | 5
  Worse by 2 points | 1 | 1 | 1
  Worse by 3 points | 0 | 0 | 1
  Worse by 4 points | 0 | 0 | 0
Statistical Analysis 1: Comparison: Vehicle Topical Solution vs ATI-50002 0.12% Topical Solution; Test type: Superiority; p = 0.602, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Vehicle Topical Solution vs ATI-50002 0.46% Topical Solution; Test type: Superiority; p = 0.643, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Change From Baseline in the Subject Global Impression of Severity of Patchy Alopecia Areata at Week 24
Description: The Subject Global Impression of Severity (SGIS) is a 5-point descriptive scale completed by subjects at Baseline, Week 4, Week 12, and Week 24 and is used to capture the subject's assessment of disease severity at a particular timepoint. Scores of 1 to 5 are assigned to responses Mild to Extremely Severe, respectively. Change status is categorized as 'Better by x points' when the score decreases from baseline by x points, and as 'Worse by x points' when the score increases by x points.
Time Frame: Baseline - Week 24
Population: Intent-to-treat population using LOCF to address missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle Topical Solution | ATI-50002 0.12% Topical Solution | ATI-50002 0.46% Topical Solution
Number analyzed (Participants) | 43 | 44 | 42
Participants
  Better by 4 points | 0 | 1 | 0
  Better by 3 points | 1 | 2 | 3
  Better by 2 points | 6 | 5 | 5
  Better by 1 point | 9 | 4 | 9
  No change | 11 | 20 | 17
  Worse by 1 point | 14 | 8 | 7
  Worse by 2 points | 2 | 4 | 1
  Worse by 3 points | 0 | 0 | 0
  Worse by 4 points | 0 | 0 | 0
Statistical Analysis 1: Comparison: Vehicle Topical Solution vs ATI-50002 0.12% Topical Solution; Test type: Superiority; p = 0.992, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Vehicle Topical Solution vs ATI-50002 0.46% Topical Solution; Test type: Superiority; p = 0.257, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: Alopecia Impact Assessment Patient Reported Outcome Change From Baseline at Week 24
Description: The Alopecia Impact Assessment (AIA) is a 13-item patient reported outcome questionnaire which measures the subject's experience with impacts related to alopecia areata in managing appearance, worry, sadness, loss of confidence, self-consciousness, embarrassment, feeling unattractive, limitation of social activities, limitation of physical activities, unwanted attention, sweat in eyes, debris in eyes, and debris in nose. The AIA was completed by subjects at Baseline, Week 4, Week 12, and Week 24 and has a recall period of "over the past seven days". An 11-point NRS with anchors "0 - Not at all [impact]" and "10 - Extremely [impact]" (e.g., "Not at all bothersome" and "Extremely bothersome"; "Not at all worried" and "Extremely worried") is utilized. The AIA produces single-item (0-10) and mean total (0-10) scores, with higher scores indicating higher levels of impact.
Time Frame: Baseline - Week 24
Population: Intent-to-treat population using LOCF to address missing data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vehicle Topical Solution | ATI-50002 0.12% Topical Solution | ATI-50002 0.46% Topical Solution
Number analyzed (Participants) | 43 | 44 | 42
score on a scale | -0.8 (2.21) | -0.8 (2.26) | -1.0 (2.30)

14. Secondary Outcome: Subject Global Impression of Treatment Satisfaction at Week 24
Description: The Subject Global Impression of Treatment Satisfaction (SGITS) is a 7-point descriptive scale completed by subjects at Week 12 and Week 24. Scale response options ranged from "1. Extremely Satisfied" to "7. Extremely Dissatisfied" and are used to capture how satisfied or dissatisfied they are with the study medication treatment received for their alopecia areata.
Time Frame: Week 24
Population: Intent-to-treat population using LOCF to address missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle Topical Solution | ATI-50002 0.12% Topical Solution | ATI-50002 0.46% Topical Solution
Number analyzed (Participants) | 38 | 41 | 38
Participants
  1. Extremely satisfied | 5 | 8 | 9
  2. Moderately satisfied | 6 | 5 | 7
  3. A little satisfied | 5 | 7 | 3
  4. Neither satisfied or dissatisfied | 5 | 8 | 6
  5. A little dissatisfied | 3 | 4 | 2
  6. Moderately dissatisfied | 5 | 3 | 4
  7. Extremely dissatisfied | 9 | 6 | 7
Statistical Analysis 1: Comparison: Vehicle Topical Solution vs ATI-50002 0.12% Topical Solution; Test type: Superiority; p = 0.374, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Vehicle Topical Solution vs ATI-50002 0.46% Topical Solution; Test type: Superiority; p = 0.253, Wilcoxon (Mann-Whitney)

15. Secondary Outcome: Change in Dermatology Life Quality Index Total Score Between Baseline and Week 24
Description: The 10 question Dermatology Life Quality Index (DLQI) questionnaire was completed by subjects at Baseline, Week 4, Week 12, and Week 24. When completing the questionnaire, subjects were instructed to think of their hair loss in place of "skin problem" and "skin" as referenced in the questionnaire. Possible summary scores could range from 0 to 30 with higher scores indicating a worse outcome.
Time Frame: Baseline - Week 24
Population: Intent-to-treat population using LOCF to address missing data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vehicle Topical Solution | ATI-50002 0.12% Topical Solution | ATI-50002 0.46% Topical Solution
Number analyzed (Participants) | 43 | 44 | 42
score on a scale | -0.5 (7.64) | -1.1 (4.07) | -2.2 (5.46)

16. Secondary Outcome: Physician Global Impression of Change at Week 24
Description: The Physician Global Impression of Change (PhGIC) is a 7-point descriptive scale completed by investigators at Week 24. Scale response options ranged from "1. Very much improved" to "7. Very much worse" and are used to capture the investigator's overall impression of change for the subject's alopecia during the treatment period.
Time Frame: Week 24
Population: Intent-to-treat population using LOCF to address missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle Topical Solution | ATI-50002 0.12% Topical Solution | ATI-50002 0.46% Topical Solution
Number analyzed (Participants) | 25 | 30 | 32
Participants
  1. Very much improved | 2 | 1 | 6
  2. Much improved | 3 | 3 | 2
  3. A little improved | 10 | 7 | 9
  4. No change | 8 | 12 | 8
  5. A little worse | 0 | 4 | 4
  6. Much worse | 1 | 1 | 1
  7. Very much worse | 1 | 2 | 2
Statistical Analysis 1: Comparison: Vehicle Topical Solution vs ATI-50002 0.12% Topical Solution; Test type: Superiority; p = 0.102, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Vehicle Topical Solution vs ATI-50002 0.46% Topical Solution; Test type: Superiority; p = 0.859, Wilcoxon (Mann-Whitney)

17. Secondary Outcome: Subject Global Impression of Change at Week 24
Description: The Subject Global Impression of Change (SGIC) is a 7-point descriptive scale completed by subjects at Week 24. Scale response options ranged from "1. Very much improved" to "7. Very much worse" and are used to capture the subject's overall impression of change for his/her alopecia during the treatment period.
Time Frame: Week 24
Population: Intent-to-treat population using LOCF to address missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle Topical Solution | ATI-50002 0.12% Topical Solution | ATI-50002 0.46% Topical Solution
Number analyzed (Participants) | 25 | 27 | 33
Participants
  1. Very much improved | 4 | 1 | 3
  2. Much improved | 2 | 4 | 6
  3. A little improved | 8 | 10 | 5
  4. No change | 3 | 4 | 8
  5. A little worse | 4 | 4 | 6
  6. Much worse | 3 | 3 | 1
  7. Very much worse | 1 | 1 | 4
Statistical Analysis 1: Comparison: Vehicle Topical Solution vs ATI-50002 0.12% Topical Solution; Test type: Superiority; p = 0.481, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Vehicle Topical Solution vs ATI-50002 0.46% Topical Solution; Test type: Superiority; p = 0.357, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Double blind period = 6 months; Open label extension period = 6 months; Reporting of non-serious AEs started with each subject's first study medication application and continued until the end of the subject's last study visit. Reporting for SAEs started when the subject signed the informed consent document and continued until the end of the subject's last visit.
Groups:
- Vehicle Topical Solution (Double Blind Period): Vehicle Topical Solution applied twice daily during the double blind period of the study.
- ATI-50002 0.12% Topical Solution (Double Blind Period): ATI-50002 0.12% Topical Solution applied twice daily during the double blind period of the study
- ATI-50002 0.46% Topical Solution (Double Blind Period): ATI-50002 0.46% Topical Solution applied twice daily during the double blind period of the study
- ATI-50002 0.46% Topical Solution (Open Label Extension Period): ATI-50002 0.46% Topical Solution applied twice daily during the open label extension period of the study
Arm/Group | Vehicle Topical Solution (Double Blind Period) | ATI-50002 0.12% Topical Solution (Double Blind Period) | ATI-50002 0.46% Topical Solution (Double Blind Period) | ATI-50002 0.46% Topical Solution (Open Label Extension Period)
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/44 | 0/42 | 0/59
Serious Adverse Events (participants affected / at risk) | 0/43 | 2/44 | 0/42 | 0/59
Other Adverse Events (participants affected / at risk) | 21/43 | 19/44 | 14/42 | 27/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vehicle Topical Solution (Double Blind Period) (N=43) | ATI-50002 0.12% Topical Solution (Double Blind Period) (N=44) | ATI-50002 0.46% Topical Solution (Double Blind Period) (N=42) | ATI-50002 0.46% Topical Solution (Open Label Extension Period) (N=59)
Application site laceration (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Polyneuropathy idiopathic progressive (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vehicle Topical Solution (Double Blind Period) (N=43) | ATI-50002 0.12% Topical Solution (Double Blind Period) (N=44) | ATI-50002 0.46% Topical Solution (Double Blind Period) (N=42) | ATI-50002 0.46% Topical Solution (Open Label Extension Period) (N=59)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0 (0) | 2 (2)
Application site exfoliation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Application site pruritis (General disorders) | 3 (3) | 1 (1) | 4 (4) | 2 (2)
Application site dermatitis (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Application site dryness (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 4 (4) | 5 (5)
Nasopharyngitis (Infections and infestations) | 2 (2) | 2 (2) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
White blood cells urine positive (Investigations) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Blood uric acid increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
High density lipoprotein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Low density lipoprotein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Lymphocyte count decreased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-04-19): https://cdn.clinicaltrials.gov/large-docs/37/NCT03354637/SAP_000.pdf
  • Study Protocol (2019-04-09): https://cdn.clinicaltrials.gov/large-docs/37/NCT03354637/Prot_001.pdf